CLINICAL TRIAL: NCT04427553
Title: Effects of Percutaneous Peripheral Nerve Stimulation on Physical Performance in Soccer Players
Brief Title: Percutaneous Peripheral Nerve Stimulation and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Full proffessor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC-UAX-02-2020
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Sports Physical Therapy
Keywords: Percutaneous Peripheral Nerve Stimulation; Performance; Soccer
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Peripheral Nerve Stimulation (Experimental): Participants assigned to this group will received two sessions (once per week) of ultrasound guided Percutaneous Peripheral Nerve Stimulation targeting the femoral nerve. We will apply a biphasic compensated electrical current at a frequency of 10 Hz, a pulse width of 240 µs and intensity allowed over a pain-free motor threshold (muscle contraction). Each participant will receive 10 repetitions of 10 seconds each one with 10 seconds rest- period between series (total treatment session 1.40 min).
  After that participants will walk during 3 minutes.
  Interventions: Device: Percutaneous Peripheral Nerve Stimulation
- Control (Placebo Comparator): Participants in the control group will walk during 5 minutes, without receiving any intervention
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Percutaneous Peripheral Nerve Stimulation — Participants assigned to this group will received two sessions (once per week) of ultrasound guided Percutaneous Peripheral Nerve Stimulation targeting the femoral nerve.
  Arms: Percutaneous Peripheral Nerve Stimulation
Other: Control Group — No intervention
  Arms: Control

SUMMARY:
Percutaneous Peripheral Nerve Stimulation is a relative new intervention applied by physical therapists. Although it has been hypothesized that this technique could improve pain and function, no studies have investigated changes in physical performance in soccer players. This study will evaluate changes in physical performance after the application of Percutaneous Peripheral Nerve Stimulation in a sample of healthy soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Semiprofessional soccer player
* No symptoms or injury in the lower extremity previous 6 months
* Training frequency of at least 3 days a week plus soccer game

Exclusion Criteria:

* fear to needles
* presence of pain or any musculoskeletal disease
* previous surgery in the lower extremity
* underlying medical conditions, e.g., diabetes, hypertension

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-04 (Actual)

PRIMARY OUTCOMES:
Changes in Contra-Movement Jump between baseline and follow-up periods | Baseline and immediately after each session and 1 month after the last treatment session
  The jump will start in an upright position with participants hands in their waists. They will perform a vertical jump after a fast down countermovement. During the knees and hips flexion, the trunk will remain the most upright as possible. The jump is measured using a Chronopump-Boscosystem DIN-A2 contact platform obtaining a jump reliable and valid height in centimeters

SECONDARY OUTCOMES:
Changes in Squat Performance Speed between baseline and follow-up periods | Baseline and immediately after each session and 1 month after the last treatment session
  The Speed4Lift device will be used. Squats will be performed using a 20kg olympic bar with two 20kg discs in each side. Participants will place the bar over their shoulders in a 90º triple-flexion position. The measurements will be performed during the concentric contraction phase of the squat

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - César Fernández-de-las-Peñas, Alcorcón, Madrid
  - César Fernández-de-las-Peñas, Alcorcón, Rest of the World